CLINICAL TRIAL: NCT05300581
Title: Determining the Feasibility of Outpatient Parenteral Antibiotic Therapy for Persons Who Inject Opioids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202110063
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observational Arm (Other): Patients with a history of injection opioid use will receive home OPAT while also receiving substance use disorder care including medications for opioid use disorder and multidisciplinary health coach and case management support.
  Interventions: Other: OPAT for PWID

INTERVENTIONS:
Other: OPAT for PWID — Observational: Patients with a history of injection opioid use will receive home OPAT while also receiving substance use disorder care including medications for opioid use disorder and multidisciplinary health coach and case management support.

SUMMARY:
Patients with a history of injection drug use are historically excluded from home outpatient parenteral antibiotic therapy programs. Recent small pilot programs have demonstrated that these patients may be safely included in home OPAT programs when they are provided with medications for opioid use disorder such as suboxone or methadone. However nothing is known about the effect of additional social support services including case management and health coach navigation on the feasibility and acceptibility of home OPAT programs for persons who inject drugs. This observational study will provide pilot data on the feasibility of such a program in anticipation of a larger scale trial.

ELIGIBILITY:
Inclusion Criteria:

* English speaking males and females
* 18-100 years of age
* Being considered for discharge from Barnes-Jewish Hospital on OPAT* (PICC/Midline only) for a serious injection related infection including; endocarditis, osteomyelitis, discitis, septic arthritis, epidural abscess, or S. aureus bacteremia. *Note that outside of this protocol patients with a history of substance use disorder are considered for discharge on OPAT to skilled nursing facilities or other health-care locations such as BJH extended care. Patients being considered for discharge on OPAT to any of these locations are eligible for inclusion.
* History of injection opioid use within the last 1 year
* Evaluated by the joint toxicology/psychiatry addiction medicine consult service during the current inpatient admission
* Started or maintained on medications for opioid use disorder (MOUD) of either methadone, buprenorphine or buprenorphine-naloxone during admission to Barnes-Jewish Hospital
* Have a scheduled follow-up for continuation of medications for opioid use disorder in place prior to discharge. For patients on methadone this should include a scheduled appointment at a methadone clinic, or for patients on buprenorphine this can include a plan for ongoing buprenorphine/ buprenorphine-naloxone based therapy at the Washington University Infectious Diseases Clinic.
* Have met with a health coach or a member of the Bridge To Health team during their inpatient hospitalization and agree to ongoing supportive counseling after discharge.
* Be willing and able to attend in-person clinic visits within 60 days post-discharge at the Washington University Infectious Diseases Clinic.
* Have a working phone number with active voicemail, running water and electricity.

Exclusion Criteria:

* Prisoner status
* Unable to provide own informed consent
* Current homelessness
* Other house-hold members reported as having active untreated substance use disorders
* Unable to attend outpatient appointments. This may include patients who are from rural areas where transportation vouchers may not provide sufficient means of making it to follow-up appointments, or other disability that would preclude transportation (paralysis, broken limbs) where the patient is unable to provide specific details as to how they would arrive at clinic appointments.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Completion of parenteral antibiotic therapy | 6 weeks patient participation
  Participants will be asked to self-report compliance to the recommended IV antibiotic therapy during a telephone survey performed at completion of antibiotic therapy.
Illicit drug use | 6 weeks patient participation
  Participants will have urine drug screens performed at clinic follow-up visit while on OPAT.

SECONDARY OUTCOMES:
Survey Completion | 3 month chart review
90-day microbiologic failure | 3 month chart review
90-day Overdose | 3 month chart review
Sample Size Estimation for Future Study | One year post-enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Laura Marks, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington Univeristy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No